CLINICAL TRIAL: NCT02422641
Title: Traditional Incision and Drainage of Cutaneous Abscess Vs. Minimally Invasive Incision and Drainage With Vessel Loop: A Randomized Controlled Trail
Brief Title: Prospective Evaluation Of High-Dose Systemic Methotrexate In Patients With Breast Cancer And Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00035551; CCCWFU 74315 (Other: WFCCC)
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer; Leptomeningeal Disease
MeSH Terms: conditions — Breast Neoplasms; Meningeal Neoplasms | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High-dose Methotrexate (8 gm/m2; HD-MTX) (Experimental): Enrolled patients will undergo treatment with HD-MTX (8 g/m2) as per current standard practice on an every 2 week schedule until disease progression or death from any cause. Treatment will be performed according to standard clinical practice. Surveillance imaging with or without cytologic evaluation will be performed as per standard clinical practice after every 2 cycles (~28 days). Treatment will continue until there is unequivocal evidence of clinical or radiographic CNS or systemic disease progression, death from any cause, or intolerance.
  Interventions: Drug: High-dose Methotrexate (8 gm/m2; HD-MTX)

INTERVENTIONS:
Drug: High-dose Methotrexate (8 gm/m2; HD-MTX) — Enrolled patients will undergo treatment with HD-MTX (8 g/m2) as per current standard practice on an every 2 week schedule until disease progression or death from any cause. Treatment will be performed according to standard clinical practice. Surveillance imaging with or without cytologic evaluation will be performed as per standard clinical practice after every 2 cycles (~28 days). Treatment will continue until there is unequivocal evidence of clinical or radiographic CNS or systemic disease progression, death from any cause, or intolerance.

SUMMARY:
Management of leptomeningeal disease (LMD) in patients with metastatic breast cancer is an area of unmet clinical need. High-dose methotrexate (HD-MTX) is known to have activity against breast cancer and in contrast to other systemic chemotherapeutics, it penetrates the blood brain barrier, targets areas of poor cerebrospinal fluid flow, may penetrate bulky leptomeningeal disease, and provide treatment to systemic disease burden. While two retrospective studies have suggested activity of HD-MTX in LMD in patients with breast cancer, no prospective data are available to inform its inclusion in treatment regimens. Thus, while HD-MTX is included in the NCCN Guidelines for LMD and while it is used to varying degrees in cancer centers across the nation, this is more representative of the lack of available therapies for LMD as opposed to strong evidence-based data. This phase II, prospective study will evaluate systemic, intravenous HD-MTX in breast cancer patients with leptomeningeal metastasis with or without brain parenchymal metastasis.

DETAILED DESCRIPTION:
BACKGROUND:

Management of LMD in patients with metastatic breast cancer is an area of unmet clinical need. Increased survival in the era of hormonal and HER2 directed therapies has further heightened the need for more effective therapies against the late complications of metastatic disease. Prognosis is dismal with median survivals ranging from 6-8 weeks in untreated patients and with little improvement having been demonstrated over the past 20 years.

Recently, there has been renewed interest in systemic chemotherapeutic options in these patients. Incorporation of systemic therapies into standard treatment algorithms has been limited as many agents have not been shown to adequately penetrate the blood brain barrier. High-dose methotrexate (HD-MTX), however, is unique in that it does penetrate the blood brain barrier. In fact, evidence suggests that it may target areas of poor cerebrospinal fluid (CSF) flow, penetrate bulk disease, and provide treatment to systemic disease burden. Methotrexate is a drug known to have activity against breast cancer and has been used in combination with cyclophosphamide and 5-fluorouracil as part of a standard adjuvant treatment regimen.

Currently, HD-MTX is included in the NCCN Guidelines for LMD and is used intermittently at Johns Hopkins and cancer centers across the nation for LMD in breast cancer. These recommendations, however, are more representative of the lack of available therapies for LMD as opposed to strong evidence-based data. Only two retrospective studies have suggested that HD-MTX may be an effective option for treating central nervous system (CNS) metastasis, both with substantial methodological limitations.

STUDY OBJECTIVE This phase II, prospective study will evaluate systemic, intravenous high-dose methotrexate (HD-MTX) in breast cancer patients with leptomeningeal metastasis (LMD). The primary objective is to determine if treatment with systemic intravenous HD-MTX will result in an overall survival (OS) exceeding 12 weeks among patients with triple negative, HER2-positive, and hormone refractory metastatic breast cancer patients with LMD with and without parenchymal brain involvement.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male and female) age >18
* Eastern Cooperative Group (ECOG) Performance Scale 0-1 (see Appendix I)
* Histologically or cytologically confirmed invasive breast cancer of the following subtype:
* TRIPLE NEGATIVE (ER-negative, PR-negative, and HER2-negative disease). Triple-negative patients will be defined per ASCO-CAP Guidelines (American Society of Clinical Oncology-College of American Pathologists).
* HER2-POSITIVE: HER2-positive patients will be defined per ASCO-CAP Guidelines.
* HORMONE REFRACTORY: Patients with ER/PR-positive disease according to ASCO-CAP guidelines above may be considered if they have disease progression after two lines of hormonal therapy (administered in the adjuvant or metastatic setting), or are deemed clinically hormone-resistant taking into consideration the rate of progression of disease or a short interval of time on first line hormonal therapy before progression. Clinically hormone-resistant patients MUST also be discussed with the investigator, co-investigator or designee in advance for approval.

NOTE: ASCO-CAP guidelines state that ER and PR assays be considered positive if there are at least 1% positive tumor nuclei in the sample on testing in the presence of expected reactivity of internal (normal epithelial elements) and external controls. HER2-positive is defined as HER2 IHC 3+, ISH ≥ 2.0, or average HER2 copy number ≥ 6.0 signals.

NOTE: A patient who has a change in receptor status (e.g. PR negative to positive) may be stratified as triple negative or hormone positive, contrary to the most recent receptor testing, for the purposes of the study, based upon the clinical course at the discretion of the Study Chair, Study co-Chair, or designee in advance for approval.

* Cytologic or unequivocal radiographic confirmation of leptomeningeal metastasis by dural puncture and/or neuroimaging with or without known brain metastasis
* Adequate organ function as follows:
* Estimated creatinine clearance >70 cc/min (calculated by Cockcroft-Gault formula)
* White blood cell counts >3000 cells/mcL
* Absolute neutrophil count >1500 cells/mcL
* Platelet count >100,000 cells/mcL
* Hematocrit >30%
* Serum bilirubin <1.5 x the ULN
* Alanine aminotransferase or aspartate aminotransferase <2.5x the ULN
* Alkaline phosphatase <2.5x the ULN or <5x the ULN if secondary to liver metastasis
* Able to provide confirmed consent

Exclusion Criteria:

* Prior allergy or adverse reaction to methotrexate
* New York Heart Association Heart Failure Class >3 (see Appendix II)
* Active diabetes insipidus
* Active mucositis
* Chemotherapy or stereotactic radiotherapy within the last 2 weeks
* Partial brain radiotherapy (i.e., less than or equal to 40% of total brain volume) within the last two weeks
* Whole brain radiotherapy within the last 6 months or partial brain radiotherapy exceeding greater than 40% of total brain volume in the last 6 months
* Prior treatment with any methotrexate containing systemic regimen within 1 year (excluding intrathecal methotrexate)
* Concurrent or planned systemic chemotherapy, radiotherapy, new hormonal or anti-HER2 directed therapy directed at management of breast cancer (existing anti-HER2 therapy can be continued as recently recommended in the National Consensus Guidelines
* Uncontrolled or progressive systemic disease or other concurrent condition which in the Investigator's opinion makes HD-MTX an undesirable treatment option for the patient or would jeopardize compliance
* Contraindication to MRI
* Use of salicylates, non-steroidal anti-inflammatory drugs, or sulfonamide medications within one week of start of methotrexate
* Pregnant women or women who are breastfeeding.
* Patients with significant visceral fluid collections including ascites, pericardial effusions, pleural effusions or others may experience delayed clearance of methotrexate because of third space accumulation which could result in methotrexate toxicity and inability to tolerate the proposed study treatment. While these are not absolute exclusions the investigators or co-investigators should be contacted to discuss possible enrollment. Patients with significant ascites defined as European Association for the Study of the Liver > grade 2, or with asymptomatic pleural effusions with an estimated size >200 mL, or with symptomatic pleural effusion of any size will be excluded.

NOTE: Systemic staging of the chest/abdomen/pelvis is required for study entry. See Sections 8.1.9. Body fluid will be assessed based on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-05; Primary Completion 2026-05 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (at 12 weeks) | 12 weeks
  The primary endpoint is survival at 12 weeks from first date of treatment. For the primary analysis, this will be dichotomized according to whether the patient achieves an OS greater than 12 weeks (i.e. survival rate). This cutoff has been selected based on reported OS data in historical controls.

SECONDARY OUTCOMES:
One year survival | 1 year
  As defined as the proportion of patients with time to death greater than 12 months from the time of first date of treatment.
Progression Free Survival | From date of first treatment to the time of systemic or neurologic progression of disease whichever occurs first, assessed up to 2 years
  Progression free survival as defined as the time from first date of treatment to the time of systemic or neurologic progression of disease whichever occurs first. Neurologic progression will be defined as the minimum of clinical or radiographic progression. Clinical neurologic progression will be defined by neurologic examination demonstrating objective, new neurologic deficit attributable to the underlying LMD. Radiographic progression (neurologic or systemic) will be defined by RECIST criteria.
Tolerability of Treatment - Number of Grade 3 or Higher Adverse Events | Up to 2 years
  Toxicity as grade 3 and higher will be tabulated by reporting period, where reporting period is defined to be the planned 14 day period between administrations of high-dose methotrexate (HD MTX).
Number of Treatment Delays | Up to 2 years
  Toxicities related to dose delays will be recorded by reporting period, where reporting period is defined to be the planned 14 day period between administrations of HD MTX. The number of times treatment is delayed divided by the number of reporting periods administered to all patients on study will be used to characterize the fraction of times treatments must be delayed.
Number of Dose Reductions | Up to 2 years
  Toxicities related to dose delays will be recorded by reporting period, where reporting period is defined to be the planned 14 day period between administrations of HD MTX. The number of times treatment is delayed divided by the number of reporting periods administered to all patients on study will be used to characterize the fraction of times treatments must be delayed.

OTHER OUTCOMES:
Treatment Cost | Up to 2 years
  As defined by the average cost per treatment course per patient.
Percentage of Cytologic Sterilization | Up to 2 years
  As defined as the percent of patients with positive baseline cytology who develop persistently negative cytology during the course of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Siteman Cancer Center- Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Comprehensive Cancer Center at Wake Forest University (CCCWFU), Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No